CLINICAL TRIAL: NCT06263478
Title: A Phase 3, Open-Label, Multicenter Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Axatilimab Monotherapy in Japanese Participants With Recurrent or Refractory Active Chronic Graft-Versus-Host Disease After at Least 2 Lines of Systemic Therapy
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Axatilimab Monotherapy in Japanese Participants With Recurrent or Refractory Active Chronic Graft-Versus-Host Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Biosciences Japan GK (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCA34176-358
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Graft-versus-host-disease
Keywords: cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Axatilimab Dose (Experimental): Axatilimab at the protocol-defined dose.
  Interventions: Drug: INCA034176

INTERVENTIONS:
Drug: INCA034176 — IV infusion
  Other Names: Axatilimab

SUMMARY:
This study will be conducted to determine the clinical efficacy of axatilimab in Japanese participants with chronic graft-versus-host disease (cGVHD).

ELIGIBILITY:
Inclusion Criteria:

* At least 6 years of age at the time of signing the ICF.
* Ability to comprehend and willingness to sign a written ICF for the study.

  • For participants 6 to 17 years old, a parent/guardian must provide consent for pediatric participants; when applicable, pediatric participants should also sign an assent form.
* Japanese participants who are allo-HSCT recipients with active, refractory, or recurrent cGVHD requiring systemic immune suppression despite at least 2 lines of prior systemic therapy.

  * Active cGVHD is defined as the presence of signs and symptoms of cGVHD per the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.
  * Refractory disease is defined as meeting any of the following criteria:

    * The development of 1 or more new sites of disease while being treated for cGVHD.
    * Progression of existing sites of disease despite at least 1 month of standard or investigational therapy for cGVHD.
    * Participants who did not achieve a response within 3 months on prior therapy for cGVHD and for whom the treating physician believes a new systemic therapy is required.
  * Recurrent cGVHD is defined as active, symptomatic disease (after an initial response to prior therapy) based on the NIH 2014 consensus criteria by organ-specific or global assessment or for which the physician believes a new line of systemic therapy is required.
* Participants may have persistent, active aGVHD and cGVHD manifestations (overlap syndrome), as defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.
* Karnofsky performance score of ≥ 60 (if aged 16 years or older); Lansky performance score of ≥ 60 (if aged younger than 16 years).
* Adequate organ and bone marrow functions evaluated during the 14 days prior to the start of study treatment.
* Creatinine clearance ≥ 30 mL/min based on the Cockcroft-Gault formula in adult participants and Schwartz formula in pediatric participants.
* Concomitant use of a systemic corticosteroid is allowed but not required. Topical and inhaled corticosteroid agents are allowed. If a participant is taking a corticosteroid, it must be a stable dose for at least 2 weeks prior to the start of study treatment.
* Concomitant use of protocol-defined immunosuppressant is allowed but not required.
* Willingness to avoid pregnancy or fathering children based on protocol-defined criteria.

Exclusion Criteria:

* Has aGVHD without manifestations of cGVHD.
* Any evidence (histologic, cytogenetic, molecular, hematologic, or mixed) of relapse of the underlying cancer or post-transplant lymphoproliferative disease at the time of screening.
* History of acute or chronic pancreatitis.
* History of myositis.
* History or other evidence of severe illness, uncontrolled infection, allergy to excipients, or any other conditions that would make the participant, in the opinion of the investigator, unsuitable for the study.
* Has acquired immunodeficiency syndrome.
* History of latent or active TB based on protocol-defined criteria.
* Active HBV or HCV infection that requires treatment, or at risk for HBV reactivation (ie, positive HBsAg).
* Pregnant or breastfeeding.
* Previous exposure to CSF-1R targeted therapies.
* Use of any agent other than corticosteroids, or the immunosuppressant for the treatment of cGVHD within 2 weeks or 5 half-lives, whichever is shorter, prior to the start of study treatment.
* Has received an investigational treatment within 28 days prior to the start of study treatment.
* Currently participating in any other interventional study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate in the First 6 Cycles | Up to Cycle 7 (Day 169)
  The overall response rate will be assessed by the number of participants with objective response by Cycle 7 (28-day cycles), Day 1, with responses defined by the 2014 NIH consensus criteria.

SECONDARY OUTCOMES:
Proportion of participants with a ≥ 7-point improvement in modified Lee symptom scale (mLSS) score | Up to 2 years
Overall Response Rate | Up to 2 years
  Defined by the 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD.
Duration of Response | Up to 2 years
  Defined as the time from initial partial response or complete response until documented progression of cGVHD, start of new therapy, or death for any reason.
Organ-specific Response Rate | Up to 2 years
  Organ-specific response is defined as the number of participants with objective response for the nine individual organs based on 2014 NIH Consensus Development Project on Criteria for Clinical Trials in cGVHD (skin, eyes, mouth, esophagus, upper gastrointestinal [GI], lower GI, liver, lungs and joints and fascia).
Percent reduction in average daily dose (or equivalent) of corticosteroids | Up to 2 years
Proportion of participants who discontinue corticosteroid use | Up to 2 years
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 years and 30 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event from the time the participant signs the informed consent form (ICF) until at least 30 days after the end of trial (EOT) or until start of new cGVHD therapy.
Change from baseline in Karnofsky/Lansky performance status | Up to 2 years and 30 days
Axatilimab pharmacokinetic (PK) in Plasma | Up to 2 years and 30 days
  Axatilimab concentration in plasma.
Number of Participants with Anti-Drug Antibody (ADA) | Up to 2 years and 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (16):
- Japan (16):
  - Fujita Health University Hospital, Aichi
  - University of Fukui Hospital, Fukui
  - Kyushu University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Hokkaido University Hospital, Hokkaido
  - Kobe City Medical Center General Hospital, Hyōgo
  - Tokai University Hospital, Kanagawa
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Tohoku University Hospital, Miyagi
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Saitama Prefectural Children'S Medical Center, Saitama-shi, Saitama,
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - National Center For Child Health and Development, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A study to evaluate the Efficacy, Safety, and Pharmacokinetics of Axatilimab Monotherapy in Japanese Participants With Recurrent or Refractory Active Chronic Graft-Versus-Host Disease — https://incyteclinicaltrials.com/studies/inca34176-358